CLINICAL TRIAL: NCT07169578
Title: A Phase III, Multicenter, Randomized, Double-Blind, Placebo-Controlled, Parallel-Group Efficacy and Safety Study of Trontinemab in Participants With Early Symptomatic Alzheimer's Disease (MCI to Mild Dementia Due to AD)
Brief Title: A Study of Trontinemab in Participants With Early Symptomatic Alzheimer's Disease
Acronym: TRONTIER 1
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: WN45443; 2024-518006-40-00 (EU CTIS Number)
Record Dates: First submitted 2025-09-10; First posted 2025-09-12 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-02

CONDITIONS: Alzheimers Disease
Keywords: Early Alzheimers Disease; Mild Cognitive Impairment; Mild Dementia
MeSH Terms: conditions — Alzheimer Disease; Cognitive Dysfunction

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Trontinemab (Experimental): Participants will receive intravenous (IV) trontinemab.
  Interventions: Drug: Trontinemab
- Placebo (Placebo Comparator): Participants will receive IV placebo.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Trontinemab — Participants will receive IV trontinemab.
  Other Names: RO7126209
  Arms: Trontinemab
Other: Placebo — Participants will receive IV placebo.
  Arms: Placebo

SUMMARY:
The purpose of this study is to assess the efficacy and safety of trontinemab in participants with early symptomatic Alzheimer's disease (AD) (mild cognitive impairment [MCI] to mild dementia due to AD).

ELIGIBILITY:
Inclusion Criteria:

* Willingness and ability to complete all aspects of the study (including MRI, clinical genotyping, and PET imaging or CSF as applicable) for the duration of the study. The participant should be capable of completing assessments either alone or with the help of the study partner
* Adequate visual and auditory acuity, in the investigator's judgment, sufficient to perform the neuropsychological testing (eyewear and hearing aids are permitted)
* Evidence of AD pathological process, as confirmed on amyloid PET scan. A CSF tau181/Aβ42 ratio may be used as an alternative option if amyloid PET is not available
* Probable AD dementia or MCI due to AD, also known as an Alzheimer's clinical syndrome clinical Stage 3 or Stage 4
* Screening MMSE score ≥ 22 and CDR-GS of 0.5 or 1.0
* Participant- and/or Informant-reported history of cognitive decline with gradual onset and progression over the last 1 year before screening
* A Repeatable Battery for the Assessment of Neuropsychological Status Delayed Memory Index (RBANS DMI) score of 85 or order
* Availability of a "study partner" as defined by the protocol

Exclusion Criteria:

* Any evidence of a condition other than AD that may affect cognition
* History or presence of clinically significant cerebrovascular disease
* History of severe, clinically significant (persistent neurologic deficit or structural brain damage) central nervous system (CNS) trauma
* History or presence of clinically significant intracranial mass
* MRI evidence of significant cerebral abnormalities or inability to tolerate MRI procedures or contraindication to MRI
* Any other medical conditions (e.g., cardiovascular, hepatic, renal disease) which are not stable and adequately controlled or which in the opinion of the investigator could affect the participant's safety in the study or interfere with the study assessments
* History of malignancy with the following exceptions: if considered to be cured; malignancies with a negligible risk of metastasis or death

Ages: 50 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 800 (Estimated)
Dates: Start 2025-09-17 (Actual); Primary Completion 2028-06-07 (Estimated); Study Completion 2028-06-07 (Estimated)

PRIMARY OUTCOMES:
Change from baseline to Week 72 in Clinical Dementia Rating, Sum of Boxes (CDR-SB) | Baseline - Week 72

SECONDARY OUTCOMES:
Change from baseline through Week 72 in Alzheimer's Disease Assessment Scale-Cognition 13 (ADAS-Cog-13) | Baseline - Week 72
Change from baseline through Week 72 in Alzheimer's Disease Cooperative Study Activities of Daily Living Inventory (ADCS-ADL) total score and instrumental score | Baseline - Week 72
Change from baseline through Week 72 in Integrated Alzheimer's Disease Rating Scale (iADRS) | Baseline - Week 72
Change from baseline through Week 72 in Mini-Mental State Examination (MMSE) | Baseline - Week 72
Change from baseline in CDR-SB | Baseline up to but excluding Week 72
Time to increase in Clinical Dementia Rating, Global Score (CDR-GS) | Baseline - Week 72
Percentage of participants with adverse events (AEs) | Baseline - Week 72
Percentage of participants with amyloid-related imaging abnormalities (ARIA) magnetic resonance imaging (MRI) findings | Baseline - Week 72
Percentage of participants with infusion-related reactions (IRR) | Baseline - Week 72
Percentage of participants with anti-drug antibodies (ADAs) to trontinemab | Baseline - Week 72
Change from baseline through Week 72 in brain amyloid load as measured by amyloid positron emission tomography (PET) scan | Baseline - Week 72
Change from baseline to Week 72 in brain tau load as measured by tau PET scan in a subset of participants | Baseline - Week 72
Change from baseline through Week 72 in cerebrospinal fluid (CSF) biomarkers of disease p-tau181, neurogranin, Aβ42 in a subset of participants | Baseline - Week 72
Change from baseline through Week 72 in blood biomarkers p-tau217, glial fibrillar acidic protein (GFAP) | Baseline - Week 72

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (108):
- United States (26):
  - Banner Sun Health Research Institute, Sun City, Arizona
  - Inglewood Clinicals, Inglewood, California
  - Irvine Center for Clinical Research, Irvine, California
  - UCSF - Memory and Aging Center, San Francisco, California
  - Syrentis Clinical Research, Santa Ana, California
  - K2 Medical Research - The Villages, Lady Lake, Florida
  - K2 Medical Research, LLC, Maitland, Florida
  - Renstar Medical Research, Ocala, Florida
  - Axiom Brain Health LLC, Tampa, Florida
  - Charter Research - Lady Lake/The Villages, The Villages, Florida
  - Alzheimer?s Research and Treatment Center, Wellington, Florida
  - Conquest Research, LLC, Winter Park, Florida
  - Accel Research Sites-NeuroStudies, Decatur, Georgia
  - Hawaii Pacific Neuroscience, Honolulu, Hawaii
  - RE:Cognition (Chicago), Chicago, Illinois
  - Boston Center for Memory, Newton, Massachusetts
  - Washington University School of Medicine, St Louis, Missouri
  - The Cognitive and Research Center of New Jersey, Ridgewood, New Jersey
  - Basil Clinical, Laurelton, New York
  - Adams Clinical Harlem, New York, New York
  - Triad Clinical Trials, Greensboro, North Carolina
  - K2 Medical Research - Nashville, Nashville, Tennessee
  - Kerwin Research Center, LLC, Dallas, Texas
  - South Texas Research Institute - Edinburg, Edinburg, Texas
  - Re:Cognition Health - Houston, Houston, Texas
  - National Clinical Research Inc.-Richmond, Richmond, Virginia
- Canada (4):
  - Richmond Clinical Trials, Richmond, British Columbia
  - Toronto Memory Program, Toronto, Ontario
  - Clinique Memoire de Montreal, Montreal, Quebec
  - Alpha Recherche Clinique, Québec
- China (21):
  - Renji Hospital Affiliated to Shanghai Jiaotong University School of Medicine, Shanghai, Shanghai Municipality
  - Peking University First Hospital, Beijing
  - Beijing Friendship Hospital Affiliated of Capital University of Medical Science, Beijing
  - The First Hospital of Jilin University, Changchun
  - West China Hospital - Sichuan University, Chengdu
  - The First Affiliated Hospital, Chongqing Medical University, Chongqing
  - Fujian Medical University Union Hospital, Fuzhou
  - Guangdong General Hospital, Guangzhou
  - The second Affiliated Hospital of Guangzhou Medical University, Guangzhou
  - Sir Run Run Shaw Hospital, School of Medicine, Zhejiang University, Hangzhou
  - The First Affiliated Hospital of Anhui Medical University, Hefei
  - Anhui Provincial Hospital, Hefei
  - Zhongda Hospital Affiliated to Southeast University, Nanjing
  - Nanjing Brain Hospital, Nanjing
  - Nanjing First Hospital, Nanjing
  - Ruijin Hospital Shanghai Jiaotong University School of Medicine, Shanghai
  - Huashan Hospital, Fudan University, Shanghai
  - Shanghai First People's Hospital, Shanghai
  - Shanghai Pudong Hospital, Shanghai
  - The Second Affiliated Hospital of Soochow University, Suzhou
  - The Affiliated Hospital of Xuzhou Medical University, Xuzhou
- France (8):
  - Hôpital Broca, Le Kremlin Bicétre Cedex
  - Hopital B Roger Salengro, Lille
  - Hôpital de la Timone, Marseille
  - Hopital Lariboisiere, Paris
  - CHU Rennes - Hopital Pontchaillou, Rennes
  - Gerontopole, Toulouse
  - CHRU - Hôpital Bretonneau, Tours
  - Hopital des Charpennes, Villeurbanne
- Germany (11):
  - Uniklinik RWTH Aachen, Aachen
  - Zentrum für klinische Forschung Dr. med. Irma Schöll, Bad Homburg
  - Klinikum Bayreuth Standort Hohe Warte Klinik fur Neurologie, Bayreuth
  - St. Josef-Hospital, Klinik für Neurologie, Bochum
  - Gesundheit Nord, Klinikum Bremen-Ost, Bremen
  - Universitätsklinikum Freiburg, Klinik für Neurologie und Neurophysiologie, Freiburg im Breisgau
  - MVZ Rheumatologie und Autoimummedizin Hamburg GmbH, Hamburg
  - Klinikum rechts der Isar der TU München, München
  - Gemeinschaftspraxis Dr. Wolfram von Pannwitz, MBA & Dr. med. Marie Perle Brinckmann, Steglitz
  - Krankenhaus der Barmherzigen Brüder Trier, Trier
  - Universitätsklinikum Ulm, Ulm
- Italy (2):
  - Fondazione Santa Lucia IRCCS, Rome, Lazio
  - IRCCS Ospedale San Raffaele, Milan, Lombardy
- Japan (10):
  - National Hospital Organization Utano National Hospital, Kyoto
  - Mishuku Hospital, Meguro-Ku
  - Mie University Hospital, Mie
  - Memory Clinic Ochanomizu, Tokyo
  - Keio University Hospital, Tokyo
  - Tokyo Metropolitan Geriatric Hospital, Tokyo
  - National Center of Neurology and Psychiatry, Tokyo
  - Federation of National Public Service Personnel Mutual Aid Associations Tachikawa Hospital, Tokyo
  - P-One Clinic, Tokyo
  - Yamagata Tokusyukai Hospital, Yamagata
- Poland (6):
  - Centrum Medyczne Neuromed Sp. z.o.o., Bydgoszcz
  - NEURO-CARE Sp. z o.o. Sp. Komandytowa, Katowice
  - ETG Neuroscience Sp. z o.o., Warsaw
  - Centrum Leczenia Zaburzen Pamieci, Warsaw
  - NZOZ WCA, Wroc?aw
  - SPSK nr 1, Zabrze
- Spain (5):
  - Hospital General De Catalunya, Sant Cugat del Vallès, Barcelona
  - Policlínica Guipuzcoa, Donostia / San Sebastian, Guipuzcoa
  - Hospital Quiron de Madrid, Pozuelo de Alarcón, Madrid
  - Hospital Universitario Reina Sofia, Córdoba
  - Hospital Universitario Dr. Peset, Valencia
- Taiwan (7):
  - Kaohsiung Medical University Hospital, Kaohsiung City
  - Taipei Medical University ?Shuang Ho Hospital, New Taipei City
  - China Medical University Hospital, North Dist.
  - Taichung Veterans General Hospital, Taichung
  - National Taiwan University Hospital, Taipei
  - Taipei Veterans General Hospital, Taipei
  - Chang Gung Medical Foundation Linkou Branch, Taoyuan
- United Kingdom (8):
  - Lynfield Mount hospital, Bradford
  - Recognition Health Bristol, Bristol
  - Surrey and Borders NHS Foundation Trust, Chertsey
  - Department of Old Age Psychiatry Kings College, London
  - RE:Cognition Health, London
  - Charing Cross Hospital, London
  - Campus for Ageing & Vitality, Newcastle
  - Tees,Esk and Wear Valleys NHS Foundation Trust, York

IPD SHARING:
Plan to Share IPD: Yes
For eligible studies, qualified researchers may request access to individual patient level clinical data. See Roche's commitment to transparency of clinical study information here: https://go.roche.com/data_sharing